CLINICAL TRIAL: NCT05766371
Title: A Phase 2 Study of Pembrolizumab Plus 177Lu-PSMA-617 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Pembrolizumab Plus 177Lu-PSMA-617 in Patients With Castration Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23551; NCI-2023-01660 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Castrate Resistant Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Prostate Cancer; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, 177Lu-PSMA-617 (Experimental): Participants will receive 400 mg of Pembrolizumab every 6 weeks and an infusion of 7.4 gigabequerel (GBq) (+/- 10%) of 177Lu-PSMA-617 on Cycle 1 Day 1 (of a 28 day cycle), and 6 weeks later, then at the first subsequent rise in PSA for up to six total doses, in the absence of unequivocal clinical progression, radiographic progression, or unacceptable toxicity, with a minimum interval of 6 weeks between doses.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda
Drug: 177Lu-PSMA-617 — Given IV
  Other Names: Lutetium-177-PSMA-617; (177Lu)-PSMA-617

SUMMARY:
This is a single-center, open-label, study of Prostate-Specific Membrane Antigen (PSMA)-targeted radionuclide therapy with 177Lu-PSMA-617 in combination with pembrolizumab in participants with metastatic castrate-resistant prostate cancer (mCRPC) who have previously progressed on at least one prior androgen pathway inhibitor (e.g., abiraterone, enzalutamide, apalutamide).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 12-month radiographic progression-free survival rate per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria in patients with mCRPC treated with pembrolizumab and 177Lu-PSMA-617.

SECONDARY OBJECTIVES:

I. To determine the median radiographic progression-free survival per RECIST v. 1.1 and PCWG3 criteria in patients with mCRPC treated with pembrolizumab and 177Lu-PSMA-617.

II. To determine the objective response rate per RECIST v. 1.1 and PCWG3 criteria in patients with mCRPC treated with pembrolizumab and 177Lu-PSMA-617.

III. To determine the median duration of objective response per RECIST v. 1.1 and PCWG3 criteria in patients with mCRPC treated with pembrolizumab and 177Lu-PSMA-617.

IV. To determine the greater than 50% decline from baseline PSA (PSA50) and greater than 90% decline from baseline PSA (PSA90) response rate by PCWG3 criteria at any time point on study, as well as individually following each dose of 177Lu-PSMA-617.

V. To determine the median time to PSA progression (TTPP) following each dose of 177Lu-PSMA-617 (e.g., TTPP-1, TTPP-2, etc.), as measured by PCWG3 criteria.

VI. To determine the median overall survival in patients with mCRPC treated with pembrolizumab and 177Lu-PSMA-617.

VII. To characterize the safety profile of the combination of pembrolizumab and 177Lu-PSMA-617 in patients with mCRPC.

EXPLORATORY OBJECTIVES:

I. To determine the lesion-specific response by baseline uptake on PSMA PET.

II. To determine the patterns of PSMA expression at the time of each TTPP event and at radiographic progression.

III. To further characterize the tumor microenvironment using Single-cell RNA sequencing (scRNA-seq) of paired metastatic tumor biopsies (a biopsy is required if there is an accessible lesion).

IV. To develop a biomarker predictive of durable response based on Cytometry by time of flight (CyTOF) profiling of whole blood samples collected at baseline and early time points on treatment.

V. To determine whether successive doses of 177Lu-PSMA-617 leads to ablation of effector T cells and up- regulation of myeloid cell states in the periphery and tumor microenvironment.

VI. To characterize participant reported outcomes using the Brief Pain Inventory and The Functional Assessment of Cancer Therapy - Prostate (FACT-P) instruments.

VII. To correlate the number of 177Lu-PSMA-617 re-priming doses and PSA progression events with radiographic rPFS.

VIII. To evaluate and compare the efficacy of 177Lu-PSMA-617 between the subgroup of participants who received a single dose of 177Lu-PSMA-617 followed by adaptive dosing, and the subgroup of participants who received two doses of 177Lu-PSMA-617 followed by adaptive dosing.

IX. To evaluate and compare efficacy between the subgroup of participants who received Schedule 1 versus Schedule 2 dosing.

X. To evaluate and compare efficacy between the subgroup of participants who have received prior taxane chemotherapy versus participants who were taxane-naïve at the time of study entry.

OUTLINE:

Participants will receive two doses of 177Lu-PSMA-617 and may continue treatment for up to a total of six total doses in the absence of unequivocal clinical progression, or unacceptable toxicity, with minimum interval of 6 weeks between doses. Participants will also receive pembrolizumab and may continue study treatment until unequivocal evidence of clinical progression or at physician's discretion based on clinical evaluation. Participants will undergo safety follow-up visits approximately 30 days and 90 days following the end of treatment visit. Participants will then be seen in clinic or contacted by telephone every 3 months to assess survival/disease/anti-cancer therapy status until death, withdrawal of consent, or the end of the study, whichever occurs first until study closure.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate adenocarcinoma that is progressive metastatic castration-resistant prostate cancer by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria at the time of study entry.
2. Male participants who are at least 18 years of age on the day of signing informed consent.
3. Castrate level of serum testosterone at study entry (< 50 ng/dL). Note: Participants without prior bilateral orchiectomy are required to remain on Luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study.
4. Prior progression on at least one second generation androgen signaling inhibitor including abiraterone, apalutamide, darolutamide, and/or enzalutamide.
5. Adverse events related to prior anti-cancer treatment (excluding LHRH analogs) must have recovered to Grade <= 1 (except for any grade alopecia and grade <= 2 neuropathy).
6. Prior radiotherapy is allowed if the last radiotherapy treatment was greater than 2 weeks from start of study treatment on cycle 1, day 1 (C1D1). Note- Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
7. At least one Prostate-Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) (PSMA PET) avid lesion on screening PSMA PET. A positive lesion is defined as uptake above background liver.
8. Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky >= 70%).
9. Demonstrates adequate organ function as defined below:

   1. Adequate bone marrow function:

      * absolute neutrophil count >=1,500/microliter (mcL)
      * platelets >=100,000/mcL
      * hemoglobin > 9.0 g/dL
   2. Adequate hepatic function:

      * total bilirubin <= 1.5 x upper limit of normal (ULN). In patients with known or suspected Gilbert's disease, direct bilirubin <= ULN
      * aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) <= 2.5 x institutional ULN (<= 5 x ULN in patients with liver metastases)
      * alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <= 2.5 x institutional upper limit of normal (<= 5 x ULN in patients with liver metastases)
   3. Adequate renal function:

      * creatinine <= 1.5 x within institutional upper limit of normal OR
      * creatinine clearance Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation or 24 hour urine collection.
10. Participants must use appropriate methods of contraception during study treatment and for at least 6 months after last study treatment. Patients who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization. Even women who use contraceptive hormones (oral, implanted, or injected), an intrauterine device, or barrier methods (diaphragms, condoms, spermicide) should be considered to be of childbearing potential. Patients who have undergone vasectomy themselves should also be considered to be of childbearing potential. Acceptable methods of contraception include continuous total abstinence, or double-barrier method of birth control (e.g., condoms used with spermicide, or condoms used with oral contraceptives). Periodic abstinence and withdrawal are not acceptable methods of contraception.
11. Participants must provide consent to comply to recommended radioprotection precautions during study.
12. Participants willing to undergo tumor biopsy and have at least one lesion safely accessible to tumor biopsy. Bone or soft tissue lesion is allowed.
13. Participants with previously treated brain metastases are eligible provided the following criteria are all met:

    1. Last treatment was > 28 days prior to C1D1.
    2. No evidence of new/progressive brain metastases is observed on magnetic resonance imaging (MRI) obtained during screening window
    3. Patient is clinically stable without requirement of steroid treatment for at least 14 days prior to first dose of study treatment on C1D1.
14. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
15. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. De novo small cell neuroendocrine prostate cancer will not be allowed due to putative lower PSMA expression in this tumor subtype. Note-Treatment-emergent small cell neuroendocrine prostate cancer detected in metastatic tumor biopsy is not excluded.
2. Soft tissue lesions (lymph nodes > 1.5 centimeter (cm) in short axis, visceral/soft tissue lesions > 1 cm) on screening Computerized tomography (CT) that are negative on PSMA PET. Note: Negative lesions on PSMA PET are defined as those with uptake below the background liver.
3. Has received other systemic anti-cancer therapies administered within 14 days, or 5 half-lives, whichever is shorter, prior to initiation of study treatment. Note: LHRH analogues are the exception.
4. Untreated brain metastases at study entry.
5. Receipt of prior PSMA-directed treatment (e.g., radiotherapy, immunotherapy, or antibody-drug conjugate).
6. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-Programmed cell death-ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX 40, CD137).
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment on C1D1. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
8. Receipt of > 2 lines of prior taxane-based chemotherapy.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g., neomercazole, carbimazole, etc.) that function to decrease the generation of thyroid hormone by a hyper-functioning thyroid gland (e.g., in Graves' disease) is not considered a form of systemic treatment of an autoimmune disease.
11. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 mg daily or other form of immunosuppressive therapy within 7 days prior to first dose of study drug.
12. Has a history of (non-infectious) ≥ grade 2 pneumonitis/interstitial lung disease that required steroids within past 2 years or has current ≥ grade 1 pneumonitis/ interstitial lung disease at the time of study enrollment.
13. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug on C1D1. Note-Administration of a killed vaccine is allowed.
14. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
15. Has clinically significant cardiovascular disease including, but not limited to:

    1. Uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure.
    2. Uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months before study entry.
    3. Clinically significant arrhythmias not controlled by medication. Note: Chronic rate controlled, or paroxysmal atrial fibrillation/flutter is not an exclusion to study participation.
16. Prior external beam radiation involving > 25 percent (%) of bone marrow or within 14 days of start of protocol therapy on C1D1.
17. Major surgery within 28 days of study treatment. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment on C1D1. Minor procedures (e.g., biopsy, cataract surgery, stent placement, endoscopy) are not considered major surgery.
18. Has an active infection requiring intravenous antibiotics within 7 days prior to C1D1.
19. Has a known history of Hepatitis B infection (defined as Hepatitis B surface antigen (HBsAg) reactive) or known active Hepatitis C virus infection (defined as (HCV RNA) [qualitative] detected, with the following exceptions:

    1. Participants who are HbsAg positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to study entry
    2. Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to study entry.
20. Has a known history of active Bacillus Tuberculosis (TB).
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. History of bleeding diathesis and currently on anti-coagulation therapy that cannot be safely discontinued for the tumor biopsy procedure.
23. Any condition that, in the opinion of the Principal Investigator, would impair the participant's ability to comply with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Median radiographic progression-free survival (rPFS) at 12 months | 12 months
  rPFS is defined as the amount of time from the initiation of study therapy and the day of first documented radiographic disease progression per RECIST version 1.1 and PCWG3 criteria. The proportion of patients without radiographic progression at 12 months from initiation of trial therapy will be reported along with the 95% confidence interval.

SECONDARY OUTCOMES:
Overall median radiographic rPFS | Up to 5 years
  rPFS is defined as the amount of time from initiation of study therapy until the participant experiences radiographic disease progression per RECIST v. 1.1 and PCWG3 criteria, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever is sooner). If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the rPFS will be censored as the last available disease assessment. Participants who discontinue treatment for clinical progression or deterioration will be included in the analysis. Results will be reported in months
Objective response rate (ORR) | Up to 10 months
  The proportion of participants treated with both 177Lu-PSMA-617 and Pembrolizumab who experience an objective response defined as a confirmed complete response (CR) or confirmed partial response (PR) per RECIST v. 1.1 and PCWG3 criteria from the initiation of trial therapy until confirmed response, disease progression, initiation of subsequent anti-cancer therapy, or participant has completed study participation (whichever occurs first). Point estimate of objective response rate will be obtained along with its 95% confidence interval.
Median duration of objective response (DOR) | Up to 10 months
  Duration of objective response is defined as the amount of time between the day of first documented response to trial therapy (confirmed CR or confirmed PR, whichever is first recorded) and subsequent disease progression (per RECIST v. 1.1 and PCWG3 criteria). Median duration of objective response will be calculated based on the using Kaplan-Meier product limit method.
Proportion of participants with 50% decline in PSA (PSA50) | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), at any point during the course of treatment.
Proportion of participants with 90% decline in PSA (PSA90) | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), at any point during the course of treatment.
Median time to PSA progression (TTPP1) following the first dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP1 is the amount of time from the date of first treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the first dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the first dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the first dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the first dose of 177Lu-PSMA-617
Median time to PSA progression (TTPP2) following the second dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP2 is the amount of time from the date of the second treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the second dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the second dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the second dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the second dose of 177Lu-PSMA-617
Median time to PSA progression (TTPP3) following the third dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP3 is the amount of time from the date of the third treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the third dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the third dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the third dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the third dose of 177Lu-PSMA-617
Median time to PSA progression (TTPP4) following the fourth dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP4 is the amount of time from the date of the fourth treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the fourth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the fourth dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the fourth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the fourth dose of 177Lu-PSMA-617
Median time to PSA progression (TTPP5) following the fifth dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP5 is the amount of time from the date of the fifth treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the fifth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the fifth dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the fifth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the fifth dose of 177Lu-PSMA-617
Median time to PSA progression (TTPP6) following the sixth dose of 177Lu-PSMA-617 | Up to 10 months
  TTPP6 is the amount of time from the date of the sixth treatment with 177Lu-PSMA-617, to the date of the first PSA level meeting the definition for PSA progression per PCWG3 criteria.
Proportion of participants with PSA50 following the sixth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 50% decline in baseline PSA (drawn at the initiation of trial therapy), following the sixth dose of 177Lu-PSMA-617
Proportion of participants with PSA90 following the sixth dose of 177Lu-PSMA-617 | Up to 10 months
  The proportion of participants who achieve greater than 90% decline in baseline PSA (drawn at the initiation of trial therapy), following the sixth dose of 177Lu-PSMA-617
Median overall survival (OS) | Up to 5 years
  OS is defined as the amount of time from the initiation of trial therapy until the date of death from any cause for all evaluable participants. Participants who discontinue from study follow up or are lost to follow up will be censored at the date of last contact. Median overall survival and 95% confidence interval will be estimated using the Kaplan-Meier method.
Percentage of participants with reported treatment-emergent adverse events | Up to 10 months
  Severity of the toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse events (including immune-related adverse events) and clinically-significant laboratory abnormalities meeting Grade 3, 4, or 5 criteria according to CTCAE, will be summarized by maximum intensity and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No